CLINICAL TRIAL: NCT00091949
Title: Insulin Resistance Intervention After Stroke (IRIS) Trial
Brief Title: Insulin Resistance Intervention After Stroke Trial
Acronym: IRIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0201013034; 5U01NS044876-10 (NIH)
Record Dates: First submitted 2004-09-20; First posted 2004-09-22 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2016-09

CONDITIONS: Stroke; Myocardial Infarction; Diabetes
Keywords: stroke; heart attack; diabetes; pioglitazone; insulin resistance
MeSH Terms: conditions — Stroke; Myocardial Infarction; Diabetes Mellitus; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Active Comparator): pioglitazone
  Interventions: Drug: pioglitazone
- Placebo (Placebo Comparator): inactive substance
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pioglitazone — a thiazolidinedione drug
  Arms: Pioglitazone
Drug: placebo — an inactive substance
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if pioglitazone is effective in preventing future strokes or heart attacks among non-diabetic persons who have had a recent ischemic stroke.

DETAILED DESCRIPTION:
Among patients throughout the world who experience a transient ischemic attack (TIA)or ischemic stroke, subsequent stroke and heart attack are major causes of death and disability. Within 4 years of the initial TIA or ischemic stroke, 16 percent of patients will have a recurrent stroke and 9 percent will have a heart attack. Prevention of further vascular events, therefore, is critically important to the health of patients with stroke.

The IRIS trial will test a new treatment strategy based on evidence linking insulin resistance to increased risk for stroke and other vascular diseases. Insulin resistance is a condition in which insulin, a normal human hormone, does not work effectively because the body is resistant to its effects. This condition can lead to diabetes and is thought to cause blood vessel disease, including stroke and heart attack, in patients with and without diabetes.

Insulin resistance affects up to 50% of stroke patients and is effectively modified with thiazolidinedione (TZD) drugs used to treat type 2 diabetes. In addition to reducing insulin resistance, these drugs have other favorable effects on blood vessels, reduce blood vessel inflammation, and potentially prevent atherosclerosis. Currently marketed TZDs include rosiglitazone and pioglitazone.

The IRIS is a clinical trial that will enroll 3936 subjects at approximately 170 hospitals in Australia, Canada, Germany, Israel, Italy, the United Kingdom (UK) and the US. After an initial screening blood test, each participant will be randomly assigned to take either pioglitazone or placebo tablets. Recruitment will be completed during 2005-2012, and all participants will be followed for a minimum of 3 years.

ELIGIBILITY:
Inclusion Criteria

1. Ages 40 years or greater at the time of randomization.
2. Ischemic stroke or TIA no less than 14 days and no more than 6 months before randomization
3. Documentation of insulin resistance as defined by a value over 3.0 on the Homeostasis Model Assessment of insulin sensitivity (HOMA).
4. Both ability and willingness to provide informed consent.
5. Presence of none of the exclusion criteria.

Exclusion Criteria

Permanent Exclusions

1. Severely disabling stroke as indicated by an inability to participate in scheduled follow-up activities.
2. Persons whose ischemic stroke or TIA was related to structural cardiac lesion, significant head trauma, proximal arterial dissection or medical instrumentation.
3. Diabetes mellitus as defined by recent use of medication for diabetes as an out-patient (*see note below) or two fasting plasma blood sugars > 126 mg/dL.
4. HgbA1c > 7.0%.
5. Irreversible medical conditions likely to affect short-term survival or ability to participate in the study protocol. These include:

   * Cancer or other chronic disease with poor prognosis (predicted survival of less than four years).
   * Severe neurologic or psychiatric disease that would complicate the evaluation of study outcomes (e.g., dementia or schizophrenia).
6. History of intolerance to any thiazolidinedione.
7. Pregnancy or desire to become pregnant.
8. Oral contraceptive use.
9. Ongoing use of oral corticosteroids.
10. History of heart failure
11. Active liver disease as defined by known liver disease accompanied by cirrhosis, significant cholestasis, portal hypertension, hepatic encephalopathy, hepatic synthetic dysfunction, or expected significant loss of liver function over the course of the study.
12. History of bladder cancer.
13. Current participation in a conflicting clinical trial. A conflicting clinical trial is defined as a trial with any of following:

    * Intervention that is known to affect the incidence of stroke or myocardial infarction.
    * Intervention that is an experimental drug.
    * Outcome that includes stroke or myocardial infarction.
    * Exclusion for participation in another trial.

Temporary Exclusions Persons with temporary exclusions may be enrolled as soon as the exclusion has resolved.

1. Alanine aminotransferase (ALT) >2.5 times the upper limit of normal.
2. Hemoglobin <8.5 g/dl.
3. Moderate or severe pitting edema of the feet or legs (IRIS grade 3 or 4).
4. Carotid surgery or carotid stenting procedure scheduled (delay randomization until 2 weeks following procedure).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3876 (Actual)
Dates: Start 2005-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter N. Kernan, M.D., Principal Investigator — Yale University
Locations (183):
- United States (99):
  - University of Alabama, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - University of Arizona, Tucson, Arizona
  - Shanti Clinical Trials (NINDS-CRC site), Colton, California
  - UCSF-Fresno, Fresno, California
  - Scripps Clinic, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California-Davis, Sacramento, California
  - University of California, San Diego, California
  - University of California, San Francisco, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - Hartford, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - National Rehabilitation Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Florida, Jacksonville, Florida
  - MIMA Century Research Associates, Melbourne, Florida
  - Pines Neurological Associates (NINDS-CRC site), Pembroke Pines, Florida
  - Floria Neurovascular Institute, Tampa, Florida
  - Cook County (Stroger) Hospital, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Ingalls Memorial Hospital (NINDS-CRC site), Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Tri-City Neruology (NINDS-CRC site), Saint Charles, Illinois
  - Indiana Medical Research, Elkhart, Indiana
  - Associates In Neurology (NINDS-CRC site), Valparaiso, Indiana
  - Iowa Health Des Moines Clinical Trials Office, Des Moines, Iowa
  - Ruan Neuroscience Center/Mercy Medical Center, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa
  - Northeast Iowa Medical Education Foundation (NINDS-CRC site), Waterloo, Iowa
  - Via Christi Regional Medical Center, Wichita, Kansas
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Penobscot Bay Neurology, Rockport, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Minneapolis Clinic of Neurology, Robbinsdale, Minnesota
  - Hattiesburg Clinic (NINDS-CRC site), Hattiesburg, Mississippi
  - St. Luke's Brain and Stroke Institute, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - St. Louis University, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Advanced Neurology Specialists, Great Falls, Montana
  - University of Nebraska, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Kessler Medical Rehab Research Corp, West Orange, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - SUNY Downstate, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - SUNY Buffalo, Buffalo, New York
  - St. Vincent's Hospital Manhattan, New York, New York
  - Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Southtowns Neurology of WNY (NINDS-CRC site), West Seneca, New York
  - Burke Medical Research Institute, White Plains, New York
  - Clinical Research of Winston-Salem, Winston-Salem, North Carolina
  - Guilford Neurologic Associates, Winston-Salem, North Carolina
  - Altru Health System, Grand Forks, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Toledo, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lankenau Institute for Medical Research, Bryn Mawr, Pennsylvania
  - Penn Stat-Hershey Medical Center (NINDS-CRC site), Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - University of Texas, Southwestern, Dallas, Texas
  - Methodist Neurological Institute, Houston, Texas
  - University of Texas, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Sentara Medical Group, Norfolk, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - Flinders Medical Centre, Bedford Park, New South Wales
  - Royal Prince Alfred, Camperstown, New South Wales
  - John Hunter Hospital (University of Newcastle), New Lambton Heights, New South Wales
  - Box Hill Hospital (Eastern Health), Box Hill, Victoria
  - Western Hospital (University of Melbourne), Footscray, Victoria
  - Austin Health (National Stroke Research Institute), Heidelberg Heights, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth, Perth, Western Australia
- Canada (12):
  - University of Alberta, Edmonton, Alberta
  - Center for Neurologic Research, Lethbridge, Alberta
  - Vancouver Island Health Research Centre, Victoria, British Columbia
  - Robarts Research Institute, London, Ontario
  - Ottawa Hospital-General Campus, Ottawa, Ontario
  - Intermountain Research Consultants, Thunder Bay, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Hôpital Charles LeMoyne, Greenfield Park, Quebec
  - McGill-Montreal General, Montreal, Quebec
  - McGill-Jewish General, Montreal, Quebec
  - Centre Hospitalier Affilie Universitaire de Quebec, Québec, Quebec
  - CHUM-Centre de recherche, Hôpital Notre-Dame, Montreal
- Germany (17):
  - Klinikum Altenburger Land, Altenburg
  - Neurologische Klinik, Bad Neustadt an der Saale
  - University Hospital-Dresden, Dresden
  - University Duesseldorf/Heinrich-Heine University, Düsseldorf
  - University of Erlangen, Erlangen
  - Alfried Krupp Hospital, Essen
  - University Hospital Frankfurt, Frankfurt
  - Freiburg University, Freiburg im Breisgau
  - Ernst-Moritz-Arndt-University Greifswald, Greifswald
  - Martin-Luther-Universitaet Halle-Wittenberg, Halle
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - University Heidelberg, Heidelberg
  - Friedrich Schiller-University Jena, Jena
  - University Hospital Mainz, Mainz
  - Klinikum der Universitat Muenchen, Munich
  - University Hospital Muenster, Münster
  - University of Ulm, Ulm
- Israel (8):
  - Soroka Medical Center, Beersheba
  - B'nai Zion Medical Center, Haifa
  - Bnai-Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Rabin Medical Center-Golda Campus, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Medical Center, Tel Aviv
- Italy (9):
  - Genoa University Hospital, Genoa
  - University of Laquila, Laquila
  - University Vita Salute San Raffaele, Milan
  - IRCCS FONdazione Istituto Neurologico C. Mondino, Pavia
  - University of Perugia, Perugia
  - University of Rome (S. Andrea Hospital), Roma
  - University of Rome La Sapienza, Rome
  - Sacred Heart Catholic University, Rome
  - Jazzolino Hospital, Vibo Valentia
- University of Puerto Rico, San Juan, Puerto Rico
- United Kingdom (29):
  - Royal Bournemouth, Bournemouth, Dorset
  - Queen Elizabeth The Queen Mother Hospital, Margate, Kent
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - Wansbeck General Hospital, Ashington, Northumberland
  - Stobhill Hospital, Glasgow, Scotland
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Southern General Hospital, Glasgow, Scotland
  - Queen Elizabeth Hospital Gateshead, Gateshead, Tyne and Wear
  - Aberdeen Royal Infirmary, Aberdeen
  - Monklands Hospital, Airdrie
  - William Harvey Hospital, Ashford
  - Royal United Hospital, Bath
  - Addenbrookes Foundation NHS Trust (Cambridge), Cambridge
  - Countess of Chester Foundation Trust, Cheshire
  - Dewsbury District Hospital, Dewsbury
  - Southend University Hospital, Essex
  - Devon PCT, Exeter
  - Royal Devon and Exeter, Exeter
  - Royal Surrey County Hospital, Guildford
  - Calderdale Royal Hospital, Halifax
  - The Royal Liverpool and Broadgreen University Hospitals, Liverpool
  - University Hospital Aintree, Liverpool
  - Kings College London, London
  - Saint Georges University of London, London
  - Luton and Dubstable Hospital, Luton
  - James Cook University Hospital, Middlesbrough
  - Newcastle upon Tyne, Newcastle upon Tyne
  - Torbay Hospital (South Devon Healthcare NHS Foundation Trust), Torquay
  - North Tyneside General Hospital, Tyne and Wear

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Viscoli CM, Brass LM, Carolei A, Conwit R, Ford GA, Furie KL, Gorman M, Guarino PD, Inzucchi SE, Lovejoy AM, Parsons MW, Peduzzi PN, Ringleb PA, Schwartz GG, Spence JD, Tanne D, Young LH, Kernan WN; IRIS Trial investigators. Pioglitazone for secondary prevention after ischemic stroke and transient ischemic attack: rationale and design of the Insulin Resistance Intervention after Stroke Trial. Am Heart J. 2014 Dec;168(6):823-9.e6. doi: 10.1016/j.ahj.2014.07.016. Epub 2014 Jul 28. PMID 25458644
- [Background] Kernan WN, Viscoli CM, Demarco D, Mendes B, Shrauger K, Schindler JL, McVeety JC, Sicklick A, Moalli D, Greco P, Bravata DM, Eisen S, Resor L, Sena K, Story D, Brass LM, Furie KL, Gutmann L, Hinnau E, Gorman M, Lovejoy AM, Inzucchi SE, Young LH, Horwitz RI; IRIS Trial Investigators. Boosting enrollment in neurology trials with Local Identification and Outreach Networks (LIONs). Neurology. 2009 Apr 14;72(15):1345-51. doi: 10.1212/WNL.0b013e3181a0fda3. PMID 19365056
- [Background] Kernan W, Viscoli C, Brass L, Amatangelo M, Birch A, Clark W, Conwit R, Furie K, Gorman M, Pesapane B, Kleindorfer D, Lovejoy A, Osborne J, Silliman S, Zweifler R, Horwitz R. Boosting enrolment in clinical trials: validation of a regional network model. Clin Trials. 2011 Oct;8(5):645-53. doi: 10.1177/1740774511414925. Epub 2011 Aug 8. PMID 21824978
- [Derived] Ridha M, Zhang C, McCullough S, Viscoli CM, Sharma R, Kamel H, Merkler AE. Silent Myocardial Infarction and Risk of Stroke Recurrence: A Post Hoc Analysis of the IRIS Trial. J Am Heart Assoc. 2025 Feb 18;14(4):e037663. doi: 10.1161/JAHA.124.037663. Epub 2025 Feb 8. PMID 39921499
- [Derived] Spence JD, Viscoli CM, Inzucchi SE, Dearborn-Tomazos J, Ford GA, Gorman M, Furie KL, Lovejoy AM, Young LH, Kernan WN; IRIS Investigators. Pioglitazone Therapy in Patients With Stroke and Prediabetes: A Post Hoc Analysis of the IRIS Randomized Clinical Trial. JAMA Neurol. 2019 May 1;76(5):526-535. doi: 10.1001/jamaneurol.2019.0079. PMID 30734043
- [Derived] Young LH, Viscoli CM, Schwartz GG, Inzucchi SE, Curtis JP, Gorman MJ, Furie KL, Conwit R, Spatz ES, Lovejoy A, Abbott JD, Jacoby DL, Kolansky DM, Ling FS, Pfau SE, Kernan WN; IRIS Investigators. Heart Failure After Ischemic Stroke or Transient Ischemic Attack in Insulin-Resistant Patients Without Diabetes Mellitus Treated With Pioglitazone. Circulation. 2018 Sep 18;138(12):1210-1220. doi: 10.1161/CIRCULATIONAHA.118.034763. PMID 29934374
- [Derived] Yaghi S, Furie KL, Viscoli CM, Kamel H, Gorman M, Dearborn J, Young LH, Inzucchi SE, Lovejoy AM, Kasner SE, Conwit R, Kernan WN; IRIS Trial Investigators. Pioglitazone Prevents Stroke in Patients With a Recent Transient Ischemic Attack or Ischemic Stroke: A Planned Secondary Analysis of the IRIS Trial (Insulin Resistance Intervention After Stroke). Circulation. 2018 Jan 30;137(5):455-463. doi: 10.1161/CIRCULATIONAHA.117.030458. Epub 2017 Oct 30. PMID 29084736
- [Derived] Kernan WN, Viscoli CM, Dearborn JL, Kent DM, Conwit R, Fayad P, Furie KL, Gorman M, Guarino PD, Inzucchi SE, Stuart A, Young LH; Insulin Resistance Intervention After Stroke (IRIS) Trial Investigators. Targeting Pioglitazone Hydrochloride Therapy After Stroke or Transient Ischemic Attack According to Pretreatment Risk for Stroke or Myocardial Infarction. JAMA Neurol. 2017 Nov 1;74(11):1319-1327. doi: 10.1001/jamaneurol.2017.2136. PMID 28975241
- [Derived] Stuart AC, Sico JJ, Viscoli CM, Tayal AH, Inzucchi SE, Ford GA, Furie KL, Cote R, Spence JD, Tanne D, Kernan WN. Taking care of volunteers in a stroke trial: a new assisted-management strategy. Stroke Vasc Neurol. 2016 Oct 25;1(3):108-114. doi: 10.1136/svn-2016-000029. eCollection 2016 Sep. PMID 28959471
- [Derived] Furie KL, Viscoli CM, Gorman M, Ford GA, Young LH, Inzucchi SE, Guarino PD, Lovejoy AM, Conwit R, Tanne D, Kernan WN; IRIS Trial Investigators. Effects of pioglitazone on cognitive function in patients with a recent ischaemic stroke or TIA: a report from the IRIS trial. J Neurol Neurosurg Psychiatry. 2018 Jan;89(1):21-27. doi: 10.1136/jnnp-2017-316361. Epub 2017 Sep 22. PMID 28939682
- [Derived] Young LH, Viscoli CM, Curtis JP, Inzucchi SE, Schwartz GG, Lovejoy AM, Furie KL, Gorman MJ, Conwit R, Abbott JD, Jacoby DL, Kolansky DM, Pfau SE, Ling FS, Kernan WN; IRIS Investigators. Cardiac Outcomes After Ischemic Stroke or Transient Ischemic Attack: Effects of Pioglitazone in Patients With Insulin Resistance Without Diabetes Mellitus. Circulation. 2017 May 16;135(20):1882-1893. doi: 10.1161/CIRCULATIONAHA.116.024863. Epub 2017 Feb 28. PMID 28246237
- [Derived] Viscoli CM, Inzucchi SE, Young LH, Insogna KL, Conwit R, Furie KL, Gorman M, Kelly MA, Lovejoy AM, Kernan WN; IRIS Trial Investigators. Pioglitazone and Risk for Bone Fracture: Safety Data From a Randomized Clinical Trial. J Clin Endocrinol Metab. 2017 Mar 1;102(3):914-922. doi: 10.1210/jc.2016-3237. PMID 27935736
- [Derived] Inzucchi SE, Viscoli CM, Young LH, Furie KL, Gorman M, Lovejoy AM, Dagogo-Jack S, Ismail-Beigi F, Korytkowski MT, Pratley RE, Schwartz GG, Kernan WN; IRIS Trial Investigators. Pioglitazone Prevents Diabetes in Patients With Insulin Resistance and Cerebrovascular Disease. Diabetes Care. 2016 Oct;39(10):1684-92. doi: 10.2337/dc16-0798. Epub 2016 Jul 27. PMID 27465265
- [Derived] Kernan WN, Viscoli CM, Furie KL, Young LH, Inzucchi SE, Gorman M, Guarino PD, Lovejoy AM, Peduzzi PN, Conwit R, Brass LM, Schwartz GG, Adams HP Jr, Berger L, Carolei A, Clark W, Coull B, Ford GA, Kleindorfer D, O'Leary JR, Parsons MW, Ringleb P, Sen S, Spence JD, Tanne D, Wang D, Winder TR; IRIS Trial Investigators. Pioglitazone after Ischemic Stroke or Transient Ischemic Attack. N Engl J Med. 2016 Apr 7;374(14):1321-31. doi: 10.1056/NEJMoa1506930. Epub 2016 Feb 17. PMID 26886418
- [Derived] Kernan WN, Inzucchi SE. Metabolic rehabilitation: science gathers to support a new intervention to prevent stroke. Stroke. 2011 Dec;42(12):3333-5. doi: 10.1161/STROKEAHA.111.632489. Epub 2011 Oct 13. No abstract available. PMID 21998067

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 1939 | 1937
Completed | 1764 | 1786
Not Completed | 175 | 151
Not completed — Withdrawal by Subject | 117 | 110
Not completed — Lost to Follow-up | 58 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 1939 | 1937 | 3876
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (10.7) | 63.5 (10.6) | 63.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 646 | 692 | 1338
  Male | 1293 | 1245 | 2538
Region of Enrollment [Number; unit: participants]
  Canada | 272 | 271 | 543
  Puerto Rico | 9 | 11 | 20
  United States | 1296 | 1276 | 2572
  United Kingdom | 123 | 133 | 256
  Italy | 22 | 26 | 48
  Israel | 90 | 88 | 178
  Australia | 53 | 55 | 108
  Germany | 74 | 77 | 151

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Fatal or Non-fatal Stroke, or Fatal or Non-fatal Myocardial Infarction
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 1939 | 1937
participants | 175 | 228
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = .0067, Regression, Cox — P-value adjusted for interim looks; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.62 to 0.93] — Pioglitazone arm compared to placebo; CI adjusted for interim looks

2. Secondary Outcome: Fatal or Non-fatal Stroke Alone
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 1939 | 1937
participants | 127 | 154
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.19, Regression, Cox — P-value adjusted for multiplicity (5 secondary outcomes); Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.61 to 1.1] — Pioglitazone arm compared to placebo; conference interval (CI) adjusted for multiplicity (5 secondary outcomes)

3. Secondary Outcome: Acute Coronary Syndrome
Description: Fatal or non-fatal acute myocardial infarction or unstable angina
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 1939 | 1937
participants | 206 | 249
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.11, Regression, Cox — P-value adjusted for multiplicity (5 secondary outcomes); Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.52 to 1.07] — Pioglitazone arm compared to placebo; CI adjusted for multiplicity (5 secondary outcomes)

4. Secondary Outcome: Development of Overt Diabetes
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 1939 | 1937
participants | 73 | 149

5. Secondary Outcome: All Cause Mortality
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 1939 | 1937
participants | 136 | 146
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.52, Regression, Cox — p-value adjusted for multiplicity (5 secondary outcomes); Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.73 to 1.17] — Pioglitazone arm compared to placebo; CI adjusted for multiplicity (5 secondary outcomes)

6. Secondary Outcome: Decline in Cognitive Status
Description: Change in modified mental status examination (3MS) score from baseline to exit. Theoretical range of 3MS scores is 0-100. Baseline scores ranged from 22-100.
Time Frame: Annual measures from baseline to exit (up to 5 years)
Population: Participants with baseline and at least 1 follow-up modified mini-mental examination score.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 1699 | 1699
units on a scale | 0.27 (0.13) | 0.29 (0.13)
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Changes in modified mini-mental examination (3MS) score from baseline (to annual scores) were analyzed using a longitudinal repeated measures mixed effects model; Test type: Superiority or Other; p = 0.88, Mixed Models Analysis; Mean Difference (Net) = -0.023, 95% CI 2-sided [-0.326 to 0.280] — Pioglitazone arm compared to placebo

7. Secondary Outcome: Composite Outcome of Fatal or Non-fatal Stroke, Fatal or Non-fatal MI or Episode of Serious Congestive Heart Failure
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 1939 | 1937
participants | 206 | 249
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.11, Regression, Cox — P-value adjusted for multiplicity (5 secondary outcomes); Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.65 to 1.05] — Pioglitazone arm compared to placebo; CI adjusted for multiplicity (5 secondary outcomes)

ADVERSE EVENTS:
Time Frame: Adverse event data collected during followup (2 to 5 years).
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 950/1939 | 987/1937
Other Adverse Events (participants affected / at risk) | 1007/1939 | 724/1937
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=1939) | Placebo (N=1937)
Hospitalization (General disorders) | 908 (1844) | 946 (2023) — Hospital stays over 24 hours during followup.
Heart failure (Cardiac disorders) | 51 (61) | 42 (55) — Heart failure resulting in hospitalization or death during followup.
Cancer (General disorders) | 133 (144) | 150 (163) — Incident cancer during followup
Bone fracture (General disorders) | 99 (178) | 62 (99) — Bone fracture requiring surgery or hospitalization during followup.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=1939) | Placebo (N=1937)
Bone fracture (General disorders) | 133 (198) | 94 (126) — Bone fracture not requiring surgery or hospitalization.
Excessive weight gain (General disorders) | 221 (892) | 88 (305) — Weight gain > 13.6 kgs from baseline at any time during followup
Edema (General disorders) | 691 (1093) | 483 (731) — New or worsening of feet or lower legs during followup
Shortness of breath (General disorders) | 342 (444) | 292 (379) — New or worse shortness of breath during followup

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No